CLINICAL TRIAL: NCT06230835
Title: Community Health Worker Led Hypertension Prevention and Control (CHPC) in Nepal: An Implementation Trial
Brief Title: Community Health Worker Led Hypertension Prevention and Control
Acronym: CHPC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Archana Shrestha, Associate Professor, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 169421-01; 1R01HL169421-01 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention of the study will be the Community Health Workers implementation strategy
  Interventions: Behavioral: Intervention Group
- Control Arm (No Intervention): Routine hypertension care

INTERVENTIONS:
Behavioral: Intervention Group — Community Health Workers (CHWs) will undergo a 4-day training program on hypertension management, including screening, counseling, medication adherence, self-care, and referrals. They will then collaborate with healthcare facilities to conduct one-day hypertension screening camps. CHWs will form self-support groups for individuals with hypertension and hold monthly meetings to discuss control strategies, review BP logs, and promote healthcare visits, including family involvement. They will also maintain regular communication with healthcare facility in-charges to ensure effective collaboration in the 'Hypertension Care Cascade Model'. No any drugs will be used in the intervention group.
  Arms: Intervention Group

SUMMARY:
With its high prevalence and concomitant increased risk of cardiovascular disease (CVD), hypertension (HTN) is a major global public health challenge. About 13.5% of premature deaths, 54% of incident stroke and 47% of incident coronary heart disease (CHD) worldwide are attributed to high blood pressure (BP). In Nepal, the prevalence of HTN among adults is 25% is similar to the global prevalence. In Nepal, however, a comparatively larger proportion of adults (44%) are unaware of their HTN status, 33% of HTN patients are receiving treatment, and only 12% of the patients have their BP under control. There are proven evidence-based interventions that have been recommended for the prevention and control of HTN including weight loss; healthy diet incorporating reduced sodium, increased fruits and vegetables, and reduced saturated fats; increased physical activity; lowered alcohol; and anti-HTN medications. Despite the availability of these proven effective lifestyle changes and low-cost anti-HTN treatment in preventing major vascular events and total mortality, these recommendations have not been translated into practice to improve population health.

In Nepal, the Package of Essential Non Communicable Diseases (PEN) Implementation Plan (2016-2020) was adopted in line with the Multi-sectoral Action Plan for the prevention and control of non communicable diseases (NCD). The PEN includes protocols to detect and manage HTN at the basic health facilities that provide primary health care incorporating all of the above-mentioned evidence-based interventions. However, our just-concluded study to evaluate the implementation of PEN in Nepal (1R21TW011718-01) demonstrated major implementation barriers at multiple levels that cannot be addressed by just health facility-based PEN: (a) Individual level: b) Interpersonal level (c) Community level (d) Organizational level.

In response to these multi-level implementation barriers, investigators propose to implement and evaluate a new task-shifting strategy to community health workers (CHW), leading to improved HTN prevention and control. Task-shifting has been proposed as a potential solution to not only address an overburdened health care system but also as a viable method for implementing primary and secondary prevention at the community-level. There is growing evidence that HTN patients can be cared for by CHW in other settings.

DETAILED DESCRIPTION:
Study Design Investigators will conduct a Hybrid type III effectiveness-implementation design focusing primarily on implementation outcomes while also collecting effectiveness outcomes as they relate to uptake or fidelity of the intervention.38 The primary implementation outcomes (aim 1) - reach, adoption, implementation and maintenance - are selected to answer the central research question of this study. Investigators will assess these outcomes in the intervention group using data from the process evaluation in intervention health facilities. To measure the effectiveness (aim2), Investigators will use a cluster-randomized design to assess effectiveness in decreasing mean systolic BP in the intervention group compared to the control group at 12 months after the intervention. Investigators will also measure cost and estimate incremental cost per participant with awareness on and control of high BP(aim 3).

Outcome Variables

Aim 1 Reach: Percentage of CHWs implementing the program will participate in at least 8 of the12 monthly meetings; Percentage of the hypertensive patients in the community are aware of their high BP status.

Adoption: Percentage of the health facilities asked to participate in adopting the program. Adoption will be a dichotomous measure --(adopted/no adopted). HF will be coded as adopting the program in CHWs completes the initial CHW training session.

Program implementation: A percentage of the health facility will implement a minimum standard to program implementation. Implementation will be a dichotomous measure (successful vs inadequate).

Maintenance: Percentage of the health facility that will implement a minimum standard to program implementation during the maintenance period. As secondary outcomes, investigators will assess the extent to which each of the individual core components were maintained, and examine the percent of health facilities implementing all core components.

Aim 2 Primary outcome: Net difference in mean systolic BP (mmHg) measured after 12 months between intervention and control group.

Aim 3 Costing: Total costs of the implementation and maintenance years by summing the costs of the individual components.

Cost-effectiveness: Investigators will estimate the cost-effectiveness in terms of incremental cost per HTN awareness, and incremental cost per BP controlled client. The primary analysis will take a financial perspective and secondary analysis will take a societal perspective.

Study Population Number of Participants Individuals with hypertension: 2432, will participate in cluster-randomized trial Community health workers: 108, will participate in focus group discussion Health workers: 84, will participate in the health worker survey Government officials: 32, will participate in key informant interview

Study setting: Investigators will include basic health facilities in Sindhupalchowk and Kavrepalanchowk districts of Bagmati province. These districts are chosen in consultation with the Province Ministry of Health (MoH) for two main reasons. First reason is the need, these are hilly districts where there are geographic challenges to deliver services through health facilities only. So, the CHW program can have the highest impact by reaching a wider community to improve HTN awareness, treatment and control. Second reason is feasibility and efficiency, these districts are the catchment areas of Dhulikhel hospital-Kathmandu University School of Medical Sciences that can directly support the program (See Letter of Support) and CHWs can refer the participants to the hospital when needed. The Provincial government has already provided permission for these health facilities to participate (See Letter of Support). In Nepal's hierarchical government structure, the provincial government commitment ensures high participation from health facilities.

Description of Intervention Local researchers will provide a 3-day training to the Community Health Workers (CHW). The CHW training will cover essential project aspects, starting with a detailed overview, including the project's introduction, aims, study area, participants, timeline, and tools. Practical sessions and role-playing exercises will be employed for the blood pressure measurement of participants, and methods for recording and reporting will be shared. The training aims to establish a foundational understanding of cardiovascular diseases, emphasizing hypertension, including its clinical features and preventive measures. The public health significance of hypertension will be underscored. The importance of diet and physical activity for the prevention of HTN will be emphasized. Specific roles and responsibilities of community health workers within the project will be highlighted. Ethical considerations, encompassing project-specific details, will be a key focus. Communication strategies for effective and culturally sensitive participant engagement will also be addressed. After receiving the training, Community Health Workers (CHW) will conduct home visits using resources from "your heart, Y: A CHW's manual for the Hispanic C" translated and adapted into Nepali and has been successfully used in the pilot Community-based intervention for blood pressure reduction in Nepal trial (COBIN) . They will visit households in their catchment area and measure BP. Each CHW will take the high BP clients (>=140/90) to the nearest health center. They will enlist the individuals with Pre Hypertension (preHTN) (preHTN and HTN and conduct three follow-up visits to these participants, every four months. In the first visit (tentative 90 minutes), CHWs will explain the purpose of the home visit and discuss HTN and its consequences. CHWs will apply inductive questioning techniques to initiate dialogue and reflection regarding lifestyle modifications and choose lifestyle goals based on PEN protocol-2, BP monitoring, and antihypertensive medication use. In subsequent visits (approximately 60 minutes), the CHWs will measure BP and address ongoing problems. The participants and family members will be engaged in a cycle of action and reflection, discussing problems faced in achieving their goals and implementing their action plans. The discussion will be tailored to the specific needs of participants and a new action plan to support will be developed as required. These interventions are realistic and feasible to implement in Nepal.

Study Visits Individuals with hypertension: intervention arm Screening and enrollment Visit-1 (Day 1-2): A trained research assistant will contact potential participants to screen for eligibility during house-to-house visits or at health facility. In this visit, that will last about 5 minutes, the research assistant will provide the purpose of the study and screening for eligibility and if the participants are interested, will provide answers to the eligibility questions. Following this, the research assistant will obtain informed consent.

Baseline survey Visit-2 (Day 1±7): Research assistants will conduct a 45-minute interview to document their socio-demographic characteristics, diet, physical activity, smoking, and alcohol history, and clinical history. The research assistants will also measure participants' height, weight, waist circumference, and blood pressure.

Intervention to intervention arm Visit 3-5 (Day 30±14, Day 120±14, Day 240±14): The intervention arm will receive a monthly session by community health workers at their home. This will be a 60-minute session, where the CHW will provide structured counseling to the participants on their lifestyle modification goals and medications; and will measure their blood pressure will record the blood pressure in a log and provide it to the research team

Endline survey Visit 6 (Day 360±14): Trained research assistants will conduct a 30-minute interview on participants' diet, physical activity, smoking, and alcohol; and will measure height, weight, waist circumference, and blood pressure.

CHWs will receive training materials covering the basics of cardiovascular diseases and emphasizing hypertension, including its clinical features and preventive measures. The manual includes counseling methods, encompassing lifestyle modification, medication, complications of HTN, preventive measures, and risk factors of HTN. The manual also includes blood pressure measurement techniques with normal and abnormal ranges. It also includes instructions to refer participants to a health facility if their blood pressure is high, with specified cut-off values.

If any participants are found to have above 180/120 mmHg, they will be referred to their primary health care (PHC) facility. The CHW or research staff will immediately call the PHC to inform about the referral.

Control arm visit:

Screening and enrollment Visit-1 (Day 1-2): A trained research assistant will contact potential participants to screen for eligibility during house-to-house visits or at health facility. In this visit, that will last about 5 minutes, the research assistant will provide the purpose of the study and screening for eligibility and if the participants are interested, will provide answers to the eligibility questions. Following this, the research assistant will obtain informed consent.

Baseline survey Visit-2 (Day 1±7): Research assistants will conduct a 45-minute interview to document their socio-demographic characteristics, diet, physical activity, smoking, and alcohol history, and clinical history. The research assistants will also measure participants' height, weight, waist circumference, and blood pressure.

Endline survey Visit-3 (Day 360±14): Trained research assistants will conduct a 30-minute interview on participants' diet, physical activity, smoking, and alcohol; and will measure height, weight, waist circumference, and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older
* have high blood pressure of 130/85 mmHg
* can provide informed consent.

Exclusion Criteria:

* severe illness requiring bed rest,
* pregnant women due to their special health needs.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2432 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reach | 1 year
  Percentage of CHWs implementing the program will participate in at least 8 of the12 monthly meetings; Percentage of the hypertensive patients in the community are aware of their high BP status.
Adoption | 1 year
  Percentage of the health facilities asked to participate in adopting the program. Adoption will be a dichotomous measure --(adopted/no adopted). Health facility (HF) will be coded as adopting the program in CHWs completes the initial CHW training session.
Program Implementation | 1 year
  A of the health facility will implement a minimum standard to program implementation. Implementation will be a dichotomous measure (successful v inadequate).
Maintenance: | 1 year
  Percentage of the health facility that will implement a minimum standard to program implementation during the maintenance period. As secondary outcomes, investigators will assess the extent to which each of the individual core components were maintained, and examine the percent of health facilities implementing all core components.
Differences in in mean systolic blood pressure | 1 year
  Net difference in mean systolic BP (mmHg) measured after 12 months between intervention and control group.
Costing | 1 year
  Total costs of the implementation and maintenance years by summing the costs of the individual components.
Cost-effectiveness | 1 year
  Investigators will estimate the cost-effectiveness in terms of incremental cost per HTN awareness, and incremental cost per BP controlled client. The primary analysis will take a financial perspective and the secondary analysis will take a societal perspective.
Difference in Body Mass Index (BMI) | 1 year
  The net difference in mean BMI was measured after 12 months between the intervention and control group. BMI will be calculated as weight in kilograms divided by hight in meters square.

CONTACTS AND LOCATIONS:
Locations (1):
- Archana Shrestha, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Background] Aryal KK, Mehata S, Neupane S, Vaidya A, Dhimal M, Dhakal P, Rana S, Bhusal CL, Lohani GR, Paulin FH, Garg RM, Guthold R, Cowan M, Riley LM, Karki KB. The Burden and Determinants of Non Communicable Diseases Risk Factors in Nepal: Findings from a Nationwide STEPS Survey. PLoS One. 2015 Aug 5;10(8):e0134834. doi: 10.1371/journal.pone.0134834. eCollection 2015. PMID 26244512
- [Background] Karmacharya BM, Koju RP, LoGerfo JP, Chan KC, Mokdad AH, Shrestha A, Sotoodehnia N, Fitzpatrick AL. Awareness, treatment and control of hypertension in Nepal: findings from the Dhulikhel Heart Study. Heart Asia. 2017 Jan 4;9(1):1-8. doi: 10.1136/heartasia-2016-010766. eCollection 2017. PMID 28123454
- [Background] Ascherio A, Rimm EB, Giovannucci EL, Colditz GA, Rosner B, Willett WC, Sacks F, Stampfer MJ. A prospective study of nutritional factors and hypertension among US men. Circulation. 1992 Nov;86(5):1475-84. doi: 10.1161/01.cir.86.5.1475. PMID 1330360
- [Background] Elliott P, Stamler J, Nichols R, Dyer AR, Stamler R, Kesteloot H, Marmot M. Intersalt revisited: further analyses of 24 hour sodium excretion and blood pressure within and across populations. Intersalt Cooperative Research Group. BMJ. 1996 May 18;312(7041):1249-53. doi: 10.1136/bmj.312.7041.1249. PMID 8634612
- [Background] He J, Tell GS, Tang YC, Mo PS, He GQ. Relation of electrolytes to blood pressure in men. The Yi people study. Hypertension. 1991 Mar;17(3):378-85. doi: 10.1161/01.hyp.17.3.378. PMID 1999367
- [Background] Cutler JA, Follmann D, Allender PS. Randomized trials of sodium reduction: an overview. Am J Clin Nutr. 1997 Feb;65(2 Suppl):643S-651S. doi: 10.1093/ajcn/65.2.643S. PMID 9022560
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Garcia-Hermoso A, Saavedra JM, Escalante Y. Effects of exercise on resting blood pressure in obese children: a meta-analysis of randomized controlled trials. Obes Rev. 2013 Nov;14(11):919-28. doi: 10.1111/obr.12054. Epub 2013 Jun 21. PMID 23786645
- [Background] Lawes CM, Vander Hoorn S, Rodgers A; International Society of Hypertension. Global burden of blood-pressure-related disease, 2001. Lancet. 2008 May 3;371(9623):1513-8. doi: 10.1016/S0140-6736(08)60655-8. PMID 18456100
- [Background] Psaty BM, Lumley T, Furberg CD, Schellenbaum G, Pahor M, Alderman MH, Weiss NS. Health outcomes associated with various antihypertensive therapies used as first-line agents: a network meta-analysis. JAMA. 2003 May 21;289(19):2534-44. doi: 10.1001/jama.289.19.2534. PMID 12759325
- [Background] Garg R, Yusuf S. Overview of randomized trials of angiotensin-converting enzyme inhibitors on mortality and morbidity in patients with heart failure. Collaborative Group on ACE Inhibitor Trials. JAMA. 1995 May 10;273(18):1450-6. PMID 7654275
- [Background] Psaty BM, Smith NL, Siscovick DS, Koepsell TD, Weiss NS, Heckbert SR, Lemaitre RN, Wagner EH, Furberg CD. Health outcomes associated with antihypertensive therapies used as first-line agents. A systematic review and meta-analysis. JAMA. 1997 Mar 5;277(9):739-45. PMID 9042847
- [Background] Parker ED, Schmitz KH, Jacobs DR Jr, Dengel DR, Schreiner PJ. Physical activity in young adults and incident hypertension over 15 years of follow-up: the CARDIA study. Am J Public Health. 2007 Apr;97(4):703-9. doi: 10.2105/AJPH.2004.055889. Epub 2007 Feb 28. PMID 17329668
- [Background] Ascherio A, Hennekens C, Willett WC, Sacks F, Rosner B, Manson J, Witteman J, Stampfer MJ. Prospective study of nutritional factors, blood pressure, and hypertension among US women. Hypertension. 1996 May;27(5):1065-72. doi: 10.1161/01.hyp.27.5.1065. PMID 8621198
- [Background] Zachariah R, Ford N, Philips M, Lynch S, Massaquoi M, Janssens V, Harries AD. Task shifting in HIV/AIDS: opportunities, challenges and proposed actions for sub-Saharan Africa. Trans R Soc Trop Med Hyg. 2009 Jun;103(6):549-58. doi: 10.1016/j.trstmh.2008.09.019. Epub 2008 Nov 6. PMID 18992905
- [Background] Jindal D, Sharma H, Gupta Y, Ajay VS, Roy A, Sharma R, Ali M, Jarhyan P, Gupta P, Srinivasapura Venkateshmurthy N, Ali MK, Narayan KMV, Prabhakaran D, Weber MB, Mohan S, Patel SA, Tandon N. Improving care for hypertension and diabetes in india by addition of clinical decision support system and task shifting in the national NCD program: I-TREC model of care. BMC Health Serv Res. 2022 May 23;22(1):688. doi: 10.1186/s12913-022-08025-y. PMID 35606762
- [Background] Labhardt ND, Balo JR, Ndam M, Grimm JJ, Manga E. Task shifting to non-physician clinicians for integrated management of hypertension and diabetes in rural Cameroon: a programme assessment at two years. BMC Health Serv Res. 2010 Dec 14;10:339. doi: 10.1186/1472-6963-10-339. PMID 21144064
- [Background] Sun Y, Mu J, Wang DW, Ouyang N, Xing L, Guo X, Zhao C, Ren G, Ye N, Zhou Y, Wang J, Li Z, Sun G, Yang R, Chen CS, He J; CRHCP Study Group. A village doctor-led multifaceted intervention for blood pressure control in rural China: an open, cluster randomised trial. Lancet. 2022 May 21;399(10339):1964-1975. doi: 10.1016/S0140-6736(22)00325-7. Epub 2022 Apr 29. PMID 35500594
- [Background] Mbuthia GW, Magutah K, Pellowski J. Approaches and outcomes of community health worker's interventions for hypertension management and control in low-income and middle-income countries: systematic review. BMJ Open. 2022 Apr 1;12(4):e053455. doi: 10.1136/bmjopen-2021-053455. PMID 35365519
- See also: Buring J, Ridker PM. Clinical Trials in Heart Disease: A Companion to Braunwald's Heart Disease. W B Saunders Company. 2004:456. — https://cir.nii.ac.jp/crid/1130000797945784832
- See also: World Health Organization, Ministry of Health and Population. Multisectoral Action Plan for the Prevention and Control of Non Communicable Diseases (2014-2020). — https://www.who.int/docs/default-source/nepal-documents/multisectoral-action-plan-for-prevention-and-control-of-ncds-(2014-2020).pdf?sfvrsn=c3fa147c_4
- See also: actors associated with Package of Essential Non-Communicable Diseases (PEN) protocol 1 Implementation in Government Health Facilities of Nepal. Nepal Health Research Council International Seminar and workshop on Public Health Action Abstract 1.3.8 — https://nhrc.gov.np/wp-content/uploads/2022/08/8th-Summit-Proceeding-Report-MD-Inner-Book.pdf
- See also: Health Authorities' Perspective on Facilitators and Barriers to Implement the Package of Essential Non-communicable Disease (PEN) in Nepal: A Qualitative Study. April 2022. Eighth National Summit of Health and Population Scientists in Nepal. — https://nhrc.gov.np/wp-content/uploads/2022/08/8th-Summit-Proceeding-Report-MD-Inner-Book.pdf
- See also: Health Service Providers' Level Facilitators and Barriers in Implementing PEN Package at Primary Healthcare Level in Nepal: A Qualitative Study. April 2022. Eighth National Summit of Health and Population Scientists in Nepal. Abstract: 2.6.13 — https://nhrc.gov.np/wp-content/uploads/2022/08/8th-Summit-Proceeding-Report-MD-Inner-Book.pdf
- See also: Patients' Perspective on Facilitators and Barriers to Utilize Non-Communicable Disease (NCD) Service at Primary Healthcare Level in Nepal: A Qualitative Study. April 2022. Eighth National Summit of Health and Population Scientists in Nepal. — https://nhrc.gov.np/wp-content/uploads/2022/08/8th-Summit-Proceeding-Report-MD-Inner-Book.pdf
- See also: Situational Analysis of Package of Essential Non-Communicable Disease (PEN) Implementation at Primary Health Care Setting in Nepal. April 2022. Eighth National Summit of Health and Population Scientists in Nepal. — https://nhrc.gov.np/wp-content/uploads/2022/08/8th-Summit-Proceeding-Report-MD-Inner-Book.pdf